CLINICAL TRIAL: NCT00873041
Title: A Randomized, Double-blind, Placebo-controlled, Phase II Study to Evaluate Efficacy and Safety of Deferasirox in Non-transfusion-dependent Thalassemia Patients With Iron Overload
Brief Title: Efficacy and Safety of Deferasirox in Non-transfusion Dependent Thalassemia Patients With Iron Overload and a One Year Open-label Extension Study
Acronym: THALASSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CICL670A2209; EudraCT 2007-007000-15 (Registry Identifier: EudraCT); NCT01185106 (obsolete NCT alias)
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-05

CONDITIONS: Non-transfusion Dependent Thalassemia
Keywords: Thalassemia; thalassemia intermedia; alpha-thalassemia; beta-thalassemia; deferasirox; iron overload; non-transfusion dependent
MeSH Terms: conditions — Thalassemia; beta-Thalassemia; alpha-Thalassemia; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 5 mg/kg/day deferasirox (Experimental): Participants received a starting dose of 5 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
  Interventions: Drug: deferasirox; Drug: placebo
- 10 mg/kg/day deferasirox (Experimental): Participants received a starting dose of 10 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
  Interventions: Drug: deferasirox; Drug: placebo
- 5 mg/kg/day placebo (Placebo Comparator): Placebo tablet matching 5 mg/kg/day orally in the morning each day for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
  Interventions: Drug: placebo
- 10 mg/kg/day placebo (Placebo Comparator): Placebo tablet matching 10 mg/kg/day orally in the morning each day for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: deferasirox — Supplied as 125 mg, 250 mg and 500 mg tablets.
  Arms: 10 mg/kg/day deferasirox; 5 mg/kg/day deferasirox
Drug: placebo — Supplied as matching 125 mg, 250 mg and 500 mg tablets.

SUMMARY:
CICL670A2209: This study will evaluate the safety and efficacy of deferasirox in non-transfusion dependent thalassemia patients with iron overload. Patients will be treated either with active treatment (deferasirox) or placebo for 12 months (core study phase). Patients who complete the core study phase will be offered to continue their study with the active treatment (deferasirox) in a 12 months extension phase. During the core and extension, the effects of treatment on iron overload in the liver will be evaluated using magnetic resonance imaging (MRI) assessments.

CICL670A2209E1: A one-year open-label extension to a randomized, double-blind, placebo-controlled, phase II study to evaluate efficacy and safety of deferasirox in non-transfusion dependent thalassemia patients with iron overload (Thalassa).

ELIGIBILITY:
Core Inclusion Criteria:

* Male or female aged ≥ 10 years with non-transfusion dependent syndromes, not requiring transfusion within 6 months prior to study start. Note: there was a local country amendment for Greece only to change the age specific inclusion criteria to ≥ 18 years old
* Liver iron concentration ≥ 5 mg/g dry weight measured by Magnetic resonance imaging (MRI) before study start
* Serum ferritin >300 ng/mL at screening

Core Exclusion Criteria:

* Hemoglobin S (HbS)-variants of thalassemia syndromes
* Anticipated regular transfusion program during the study. Patients having a sporadic transfusion (e.g. in case of infection) throughout the study course will not be excluded
* Any blood transfusion 6 months prior to study start
* Creatinine clearance ≤ 60 mL/min at screening
* Serum creatinine above the upper limit of normal at both screening visits
* Significant proteinuria as indicated by a urine protein/urine creatinine ratio > 1.0 mg/mg
* Alanine aminotransferase (ALT) of > 5 x the upper limit of normal at both screening visits
* Concomitant therapy with hydroxyurea, erythropoietin, butyrate
* History of deferasirox treatment
* Pediatric patients: a patient's weight of below 20 kg

Extension Inclusion Criteria:

* Patients who completed the core CICL670A2209 clinical trial
* Written informed consent obtained prior entry to one year extension study CICL670A2209

Extension Exclusion Criteria:

* Patients with a continuous increase in serum creatinine ≥ 33% above the baseline value and > ULN who did not improve after drug interruption or dose reduction in the core study
* Patients with a continuous increase in ALT greater than 2 times the baseline value and > 5 times ULN who did not improve after drug interruption or dose reduction in the core study
* Patients with progressive proteinuria, as assessed by the investigator, who did not improve after drug interruption or dose reduction in the core study
* Significant medical condition interfering with the ability to partake in this study (e.g.systemic uncontrolled hypertension, unstable cardiac disease not controlled by standard medical therapy, systemic disease (cardiovascular, renal, hepatic, etc.)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (3):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's Memorial Hospital/Division of Hematology/Oncology, Chicago, Illinois
  - New York Presbyterian Hospital/Weill Medical College of Cornell University, New York, New York
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Italy (5):
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Rome
- Novartis Investigative Site, Beirut, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Ampang Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Taipei, Taiwan
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Taher AT, Porter JB, Viprakasit V, Kattamis A, Chuncharunee S, Sutcharitchan P, Siritanaratkul N, Origa R, Karakas Z, Habr D, Zhu Z, Cappellini MD. Defining serum ferritin thresholds to predict clinically relevant liver iron concentrations for guiding deferasirox therapy when MRI is unavailable in patients with non-transfusion-dependent thalassaemia. Br J Haematol. 2015 Jan;168(2):284-90. doi: 10.1111/bjh.13119. Epub 2014 Sep 12. PMID 25212456
- [Derived] Taher AT, Porter JB, Viprakasit V, Kattamis A, Chuncharunee S, Sutcharitchan P, Siritanaratkul N, Galanello R, Karakas Z, Lawniczek T, Habr D, Ros J, Zhang Y, Cappellini MD. Deferasirox demonstrates a dose-dependent reduction in liver iron concentration and consistent efficacy across subgroups of non-transfusion-dependent thalassemia patients. Am J Hematol. 2013 Jun;88(6):503-6. doi: 10.1002/ajh.23445. Epub 2013 May 13. PMID 23553596
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 4 week screening period to determine eligibility prior to randomization.
Groups:
- Placebo/Deferasirox: Placebo tablet matching 5 mg/kg/day or 10 mg/kg/day orally in the morning each day for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
Period: Core Study
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo/Deferasirox
Started | 55 | 55 | 56
Completed | 48 | 49 | 51
Not Completed | 7 | 6 | 5
Not completed — Adverse Event | 2 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Abnormal laboratory value | 0 | 0 | 1
Not completed — Protocol deviation | 1 | 0 | 1
Period: Extension Study
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo/Deferasirox
Started | 41 | 44 | 48
Completed | 40 | 44 | 46
Not Completed | 1 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Administrative reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo tablet matching 5 mg/kg/day or 10 mg/kg/day orally in the morning each day for 52 weeks. Participants received a starting dose of 5 or 10 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo | Total
Number analyzed (Participants) | 55 | 55 | 56 | 166
Age, Customized [Number; unit: Participants]
  <18 years | 6 | 7 | 8 | 21
  Between 18 and 65 years | 49 | 47 | 48 | 144
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 25 | 77
  Male | 29 | 29 | 31 | 89

OUTCOME MEASURES:

1. Secondary Outcome: Core Study: Change in Liver Iron Concentration (LIC) From Baseline to Week 24
Description: LIC was measured by magnetic resonance imaging technique at baseline and Week 24. Estimates were obtained from an Analysis of Covariance (ANCOVA) model for change in LIC between baseline and Week 24 with treatment as factor and baseline LIC as covariate.
Time Frame: Baseline, Week 24
Population: Full Analysis Set. The last available post-baseline LIC was carried forward if no LIC value was available at Week 24. Only patients with both baseline and at least one post-baseline value were included for this analysis.
Measure: Least Squares Mean (Standard Error); unit: mg iron (Fe)/g dry weight (dw)
Groups:
- 5 mg/kg/Day Deferasirox: Participants received a starting dose of 5 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
- 10 mg/kg/Day Deferasirox: Participants received a starting dose of 10 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
- Placebo: Placebo tablet matching 5 mg/kg/day or 10 mg/kg/day orally in the morning each day for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 49 | 48 | 51
mg iron (Fe)/g dry weight (dw) | -0.87 (0.448) | -0.90 (0.450) | -0.24 (0.439)

2. Secondary Outcome: Core Study: Change in Serum Ferritin Between Baseline and Fourth Quarter
Description: Baseline serum ferritin average was the average of all available ferritin values from screening to last sample prior to the first intake of study drug.
  Fourth quarter serum ferritin average was the average of all serum ferritin values obtained within days 286- End of Study.
  Change from baseline: fourth quarter serum ferritin average - baseline serum ferritin average.
Time Frame: Baseline, (Day 286 to End of Study [Day 365])
Population: Full Analysis set (all randomized patients). Only participants with both baseline and post-baseline values are included in analyses. If serum ferritin was missing during the fourth quarter, the last available average of serum ferritin per quarter was used for the calculation of the change from baseline.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 51 | 50 | 53
μg/L | -130.47 (260.555) | -249.16 (389.356) | 128.63 (249.689)

3. Secondary Outcome: Core Study: Change in Serum Ferritin Between Baseline and Second Quarter
Description: Baseline serum ferritin average was the average of all available ferritin values from screening to last sample prior to the first intake of study drug.
  Second quarter serum ferritin average was the average of all serum ferritin values obtained within days 106-195.
  Change from baseline: second quarter serum ferritin average - baseline serum ferritin average.
Time Frame: Baseline, (Day 106 to Day 195)
Population: Full Analysis set (all randomized patients). Only participants with both baseline and post-baseline values are included in analyses. If serum ferritin was missing during the second quarter, the last available average of serum ferritin per quarter was used for the calculation of the change from baseline.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 52 | 54 | 56
μg/L | 8.20 (244.443) | -17.75 (368.812) | 106.45 (330.217)

4. Secondary Outcome: Core Study: Percentage of Participants With Adverse Events Graded Mild, Moderate and Severe
Description: Percentage of Participants with Mild, Moderate and Severe adverse events (AE) any primary system organ class regardless of study drug relationship. A patient with multiple occurrences of an AE is counted only once in the AE category for that treatment. A patient with multiple severity ratings for an AE while on a treatment is only counted once under the maximum rating.
Time Frame: 52 Weeks
Population: Safety Analysis Set included all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 55 | 55 | 56
Percentage of participants
  Mild | 36.4 | 43.6 | 42.9
  Moderate | 27.3 | 16.4 | 21.4
  Severe | 12.7 | 18.2 | 16.1

5. Secondary Outcome: Core Study: Change in Liver Iron Concentration (LIC) From Baseline At Week 24 and Week 52 in Patients With Dose Increases After Week 24
Description: LIC was measured by magnetic resonance imaging technique at baseline, Week 24 and Week 52. Dose Doubling (Dose Increases) began at Week 24.
Time Frame: Baseline, Week 24, Week 52
Population: Full Analysis Set. The last available post-baseline LIC was carried forward if no LIC value was available at Week 24 and Week 52. Only patients with dose increases after week 24, with both baseline and at least one post-baseline value were included for this analysis.
Measure: Mean (Standard Deviation); unit: mg iron (Fe)/g dry weight (dw)
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 26 | 25 | 30
mg iron (Fe)/g dry weight (dw)
  Change from baseline at Week 24 (n=26,24,30) | 0.56 (2.992) | 0.69 (3.131) | 0.94 (2.693)
  Change from baseline at Week 52 | -1.82 (3.101) | -4.02 (4.849) | 0.62 (4.128)

6. Secondary Outcome: Core Study: Correlation Between Serum Ferritin and LIC (Liver Iron Concentration)
Description: The correlation between serum ferritin and LIC was investigated using a scatter plot with a regression line for the following cases:
  * Baseline serum ferritin versus baseline LIC
  * Serum ferritin difference from baseline at fourth quarter versus difference from baseline in LIC at Week 52.
  A value of 1.0 indicates a perfect correlation.
Time Frame: Baseline, 52 weeks
Population: Participants from the Full Analysis Set (all randomized participants).
Measure: Number; unit: Correlation coefficient
Groups:
- All Randomized Participants: Participants received a starting dose of 5 mg/kg/day or 10 mg/kg/day deferasirox tablets or matching placebo orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 165
Correlation coefficient
  Baseline | 0.653
  Week 52 (n=134) | 0.609

7. Secondary Outcome: Core Study: Change From Baseline in Hemoglobin at Month 12
Description: Blood was collected for Hemoglobin at baseline and Month 12. Change from baseline= Month 12 hemoglobin - baseline hemoglobin.
Time Frame: Baseline, Month 12
Population: Full Analysis Set (all randomized participants). Only patients with a value both at baseline and at considered timepoint are included in analyses.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 47 | 48 | 49
g/L | -1.8 (5.45) | -0.7 (6.27) | -2.8 (7.31)

8. Secondary Outcome: Core Study: Change From Baseline in Transferrin Saturation at Month 12
Description: Blood was collected for transferrin saturation at Baseline and Month 12. Change from baseline= Month 12 transferrin saturation - baseline transferrin saturation.
Time Frame: Baseline, Month 12
Population: Full Analysis Set (all randomized patients). Only patients with a value both at baseline and at considered timepoint are included in the analyses.
Measure: Mean (Standard Deviation); unit: Percent saturation
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 47 | 47 | 47
Percent saturation | -3.79 (14.234) | -3.64 (22.443) | 3.37 (10.083)

9. Secondary Outcome: Core Study: Change in Liver Iron Concentration (LIC) in Placebo Patients From Baseline to Week 52
Description: LIC was measured by magnetic resonance imaging technique at baseline and Week 52. The change in liver iron concentration for participants in the placebo arm was used to assess the iron accumulation rate.
Time Frame: Baseline, Week 52
Population: Safety Analysis Set. The last available post-baseline LIC was carried forward if no LIC value was available at Week 52. Only patients with both baseline and at least one post-baseline value were included for this analysis.
Measure: Mean (Standard Deviation); unit: mg iron (Fe)/g dry weight (dw)
Arm/Group | Placebo
Number analyzed (Participants) | 54
mg iron (Fe)/g dry weight (dw) | 0.26 (3.501)

10. Secondary Outcome: Core Study: Percentage of Participants With Notable Abnormal Post-baseline Laboratory Results
Description: The percentage of participants with notable laboratory results:
  Platelet count: (<100 x 10^9/L)
  Absolute neutrophils: (<1.5 x 10^9/L)
  Alanine aminotransferase (ALT): (>5 x Upper limit normal (ULN) and >2 x baseline).
  Aspartate aminotransferase (AST): (>5 x ULN and >2 x baseline)
  Serum creatinine: (>33% increase from baseline and >ULN at ≥2 consecutive post-baseline values) Creatinine clearance: (<60 mL/min at ≥2 consecutive post-baseline values)
  Urinary protein/creatinine ratio: (≥ 1.0 mg/mg at ≥2 consecutive post-baseline values)
Time Frame: 52 Weeks
Population: Safety Set included all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Placebo tablet matching 5 mg/kg/day or 10 mg/kg/day orally in the morning each day for 52 weeks. Participants received a starting dose of 5 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation.
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 55 | 55 | 56
Percentage of participants
  Platelet count | 5.5 | 5.5 | 10.7
  Absolute neutrophils | 5.5 | 3.6 | 5.4
  ALT | 0 | 0 | 1.8
  AST | 0 | 1.8 | 1.8
  Serum creatinine | 0 | 5.5 | 0
  Creatinine clearance | 1.8 | 1.8 | 0
  Urinary protein/creatinine ratio | 1.8 | 0 | 0

11. Primary Outcome: Core Study: Change in Liver Iron Concentration (LIC) From Baseline to Week 52
Description: LIC was measured by magnetic resonance imaging technique at baseline and Week 52. Estimates were obtained from an Analysis of Covariance (ANCOVA) model for change in LIC between baseline and Week 52 with treatment as factor and baseline LIC as covariate.
Time Frame: Baseline, Week 52
Population: Full Analysis Set. The last available post-baseline LIC was carried forward if no LIC value was available at Week 52. Only patients with both baseline and at least one post-baseline value were included for this analysis.
Measure: Least Squares Mean (Standard Error); unit: mg iron (Fe)/g dry weight (dw)
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 51 | 54 | 54
mg iron (Fe)/g dry weight (dw) | -1.95 (0.500) | -3.80 (0.484) | 0.38 (0.486)

12. Secondary Outcome: Core Study: Percentage of Participants With Notably Abnormal Post-baseline Systolic Blood Pressure
Description: Systolic blood pressure was measured at each visit after the patient rested in the sitting position for at least 3 minutes.
  A Notably Abnormal Systolic Blood Pressure was defined as a measurement in one of the following two categories:
  High: ≥180 with an increase from baseline ≥20 mmHg
  Low: ≤90 with a decrease from baseline ≥20 mmHg
Time Frame: Baseline, 52 Weeks
Population: Safety Set includes all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 55 | 55 | 56
Percentage of participants
  High | 0.0 | 0.0 | 1.8
  Low | 10.9 | 5.5 | 16.1

13. Secondary Outcome: Core Study: Percentage of Participants With Notably Abnormal Post-baseline Diastolic Blood Pressure
Description: Diastolic blood pressure was measured at each visit after the patient rested in the sitting position for at least 3 minutes.
  A Notably Abnormal Diastolic Blood Pressure was defined as a measurement in one of the following two categories:
  High: ≥105 with an increase from baseline ≥15 mmHg
  Low: ≤50 with a decrease from baseline ≥15 mmHg
Time Frame: Baseline, 52 Weeks
Population: Safety Set includes all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 55 | 55 | 56
Percentage of participants
  High | 0.0 | 0.0 | 0.0
  Low | 14.5 | 10.9 | 14.3

14. Secondary Outcome: Core Study: Percentage of Participants With Notably Abnormal Post-baseline Pulse Rate
Description: Pulse Rate was measured at each visit.
  A Notably Abnormal Pulse Rate was defined as a measurement in one of the following two categories:
  High: ≥120 with an increase from baseline ≥15 beats per minute (bpm)
  Low: ≤50 with a decrease from baseline ≥15 bpm
Time Frame: Baseline, 52 Weeks
Population: Safety Set includes all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg/kg/Day Deferasirox | 10 mg/kg/Day Deferasirox | Placebo
Number analyzed (Participants) | 55 | 55 | 56
Percentage of participants
  High | 1.8 | 0.0 | 3.6
  Low | 0.0 | 1.8 | 0.0

15. Secondary Outcome: Extension Study: Absolute Change in Serum Ferritin From Baseline to Eighth Quarter
Description: Blood was collected for serum ferritin at Core Baseline and monthly during the Eighth quarter of the Extension Study. Absolute change from Baseline: quarterly average - baseline average. A negative change from baseline indicated improvement.
Time Frame: Core Baseline, Eighth Quarter (last 3 months of the study)
Population: Full Analysis Set included all randomized participants. Only patients with a value both at baseline and at considered time point are included.
Measure: Mean (Standard Deviation); unit: micrograms/liter
Groups:
- Deferasirox: Participants received a starting dose of 5 mg/kg/day or 10 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
Arm/Group | Deferasirox | Placebo/Deferasirox
Number analyzed (Participants) | 84 | 46
micrograms/liter | -565.9 (504.25) | -504.3 (770.60)

16. Primary Outcome: Extension Study: Percentage of Participants Reaching a Liver Iron Concentration (LIC) < 5 mg Fe/g dw From Core Baseline to End of Extension Study
Description: Liver iron concentration was measured at Core Baseline and at the end of the Extension Study. Magnetic Resonance Imaging (MRI) scans were analyzed at a central laboratory to determine the LIC value. The percentage of participants with LIC < 5 mgFe/g dw (milligram iron/gram dry weight) change from Baseline at the end of the Extension Study is reported.
Time Frame: Core Baseline to End of Extension Study (up to 24 months)
Population: Full Analysis consisted of all randomized participants. Patients with post-baseline LIC satisfying criterion at any time during the study are counted as responder. Patients with no baseline LIC or without any post-baseline LIC measurements will be assumed as non-responder.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Deferasirox | Placebo/Deferasirox
Number analyzed (Participants) | 110 | 56
Percentage of participants | 39.1 [30.5 to 48.4] | 37.5 [26.0 to 56.0]

17. Secondary Outcome: Extension Study: Change in Liver Iron Concentration (LIC) From Baseline at Month 24
Description: LIC was measured by magnetic resonance imaging technique at Baseline and Month 24. A negative change from baseline indicated improvement.
Time Frame: Core Baseline, Month 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg iron (Fe)/g dry weight (dw)
Arm/Group | Deferasirox | Placebo/Deferasirox
Number analyzed (Participants) | 84 | 46
mg iron (Fe)/g dry weight (dw) | -7.1 (5.3) | -6.7 (6.67)

18. Secondary Outcome: Extension Study: Correlation Between Serum Ferritin and LIC (Liver Iron Concentration)
Description: The correlation between serum ferritin and LIC was investigated using a scatter plot with a regression line for serum ferritin difference from Baseline at Month 24 versus LIC difference from Baseline at Month 24.
  A value of 1.0 indicates a perfect correlation.
Time Frame: Core Baseline, Month 24
Population: Participants from the Extension Full Analysis Set (all randomized participants)in the Extension Study with data available for analysis.
Measure: Number; unit: Correlation coefficient
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 129
Correlation coefficient | 0.735

19. Secondary Outcome: Extension Study: Change From Baseline in Hemoglobin at Month 24
Description: Blood was collected for Hemoglobin at Baseline and Month 24. Change from Baseline= Month 24 hemoglobin - Baseline hemoglobin.
Time Frame: Core Baseline, Month 24
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: g/L
Groups:
- Deferasirox: Participants received a starting dose of 5 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
Arm/Group | Deferasirox | Placebo/Deferasirox
Number analyzed (Participants) | 59 | 29
g/L | -2.6 (6.07) [-4.19 to -1.03] | -3.1 (9.48) [-6.73 to 0.48]

20. Secondary Outcome: Extension Study: Change From Baseline in Transferrin Saturation at Month 24
Description: Blood was collected for transferrin saturation at Baseline and Month 24. Change from baseline= Month 24 transferrin saturation - baseline transferrin saturation.
Time Frame: Core Baseline, Month 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percent saturation
Arm/Group | Deferasirox | Placebo/Deferasirox
Number analyzed (Participants) | 66 | 33
Percent saturation | -5.01 (24.36) [-11.00 to 0.98] | 1.35 (13.01) [-3.26 to 5.97]

ADVERSE EVENTS:
Groups:
- Deferasirox 5 mg/kg/Day: Participants received a starting dose of 5 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
- Deferasirox 10 mg/kg/Day: Participants received a starting dose of 10 mg/kg/day deferasirox tablets orally each day in the morning for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
- Placebo/Deferasirox Any Dose: Placebo tablet matching 5 mg/kg/day or 10 mg/kg/day orally in the morning each day for 52 weeks. After 24 weeks of treatment Liver Iron Concentration (LIC) was assessed. Based on the LIC and change from baseline in LIC participants were eligible for dose escalation. In the Extension Study participants received deferasirox once daily (dose based on LIC) for 52 weeks.
Arm/Group | Deferasirox 5 mg/kg/Day | Deferasirox 10 mg/kg/Day | Placebo/Deferasirox Any Dose
Serious Adverse Events (participants affected / at risk) | 11/55 | 12/55 | 16/56
Other Adverse Events (participants affected / at risk) | 37/55 | 45/55 | 48/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox 5 mg/kg/Day (N=55) | Deferasirox 10 mg/kg/Day (N=55) | Placebo/Deferasirox Any Dose (N=56)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Babesiosis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 4 | 2
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
C-reactive protein (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox 5 mg/kg/Day (N=55) | Deferasirox 10 mg/kg/Day (N=55) | Placebo/Deferasirox Any Dose (N=56)
Anaemia (Blood and lymphatic system disorders) | 6 | 4 | 3
Conjunctivitis (Eye disorders) | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 4 | 9 | 7
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 8 | 7 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 3 | 4
Gastritis (Gastrointestinal disorders) | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 5 | 9 | 12
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3 | 8
Asthenia (General disorders) | 2 | 1 | 3
Fatigue (General disorders) | 3 | 7 | 6
Oedema peripheral (General disorders) | 1 | 1 | 4
Pain (General disorders) | 3 | 0 | 1
Pyrexia (General disorders) | 10 | 5 | 15
Gastroenteritis (Infections and infestations) | 3 | 5 | 4
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 2
Influenza (Infections and infestations) | 4 | 6 | 5
Nasopharyngitis (Infections and infestations) | 6 | 5 | 6
Pharyngitis (Infections and infestations) | 6 | 2 | 2
Rhinitis (Infections and infestations) | 2 | 5 | 3
Tonsillitis (Infections and infestations) | 5 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 14 | 14
Viral infection (Infections and infestations) | 2 | 0 | 4
Blood creatinine increased (Investigations) | 1 | 3 | 2
Heart rate increased (Investigations) | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Dizziness (Nervous system disorders) | 4 | 0 | 1
Headache (Nervous system disorders) | 3 | 11 | 12
Insomnia (Psychiatric disorders) | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.